CLINICAL TRIAL: NCT02953626
Title: Mother Matters: Pilot Randomized Waitlist Controlled Trial of an Online Postpartum Mental Health Support Group
Brief Title: Mother Matters Online Postpartum Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Collaborators: Centre for Addiction and Mental Health (Other); Sunnybrook Health Sciences Centre (Other); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0032-B
Record Dates: First submitted 2016-06-13; First posted 2016-11-03 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Depression
Keywords: pilot RCT; waitlist-controlled RCT; postpartum depression
MeSH Terms: conditions — Depression; Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Treatment Condition (ITC) (Experimental): Mother Matters Online Postpartum Support Group. Participants will be assigned to begin immediately after randomization.
  Interventions: Behavioral: Mother Matters Online Postpartum Support Group
- Waitlist Control Condition (WLC) (No Intervention): Mother Matters Online Postpartum Support Group. Participants will receive the intervention after the Immediate Treatment Condition group completes the intervention, and after follow-up data are collected from both groups.

INTERVENTIONS:
Behavioral: Mother Matters Online Postpartum Support Group — Mother Matters is a 10-week online support group for women with postpartum depression. It involves: 1) A private, online forum that can be accessed by participants 24-hours per day. During regular business hours (9:00 am to 5:00 pm on weekdays) it is moderated by a psychotherapist, and there is a weekly moderated "live" chat hour; 2) Weekly topics with readings are provided with questions to prompt discussion on the online forum. Topics incorporate symptom management (i.e. Interpersonal Therapy, Cognitive Behavioural Therapy) and affect regulation strategies (i.e. Mindfulness, DBT) with a supportive counselling approach. External resources related to each week's topic, are also shared.
  Arms: Immediate Treatment Condition (ITC)

SUMMARY:
Postpartum depression is common, yet only 20% of women seek treatment. Online support groups are a potential means of providing accessible mental health care during this time. Mother Matters is a 10-week online psychotherapy group for women with postpartum depression & anxiety. The investigators aim to conduct a pilot RCT to demonstrate the feasibility of proceeding to a large-scale RCT evaluation of the Mother Matters intervention.

DETAILED DESCRIPTION:
The postpartum period is a particularly vulnerable time for the development of mental health concerns; postpartum depression (i.e. depression with onset between 0-12 months postpartum) affects approximately 13% of mothers in Canada. There are serious negative consequences to both mother and child during this period, yet only 20% of women seek treatment, citing significant systematic and personal barriers. Online support groups have been identified as a potential means of providing accessible mental health care during this time. Mother Matters is a 10-week online support group for women with postpartum depression and anxiety, run trained psychotherapists in the Reproductive Life Stages (RLS) program at Women's College Hospital in Toronto, Ontario. Mother Matters was designed to address barriers related to accessing postpartum mental health services: it can be accessed anywhere (online group), at any time (available 24/7), and with anonymity (to address the barrier of shame/stigma). The overall objective of the current pilot RCT is to determine the feasibility of conducting a large randomized controlled trial to evaluate the efficacy of the group, comparing outcomes among those with and without access to the program.

ELIGIBILITY:
Inclusion Criteria

The specific inclusion criteria for this group are women who are:

1. Mothers of a baby/babies between 0 and 12 months old at enrollment, and
2. Over 18 years old, and
3. Have an Edinburgh Postnatal Depression Scale (EPDS) score of >9, and
4. Reside in Ontario.

Exclusion Criteria

Women will not be eligible to participate in the study if they are:

1. Experiencing active suicidal ideation, or
2. Have active substance use, mania or psychosis, or
3. Unable to access the internet, or
4. Unable to participate in English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-05; Primary Completion 2017-03 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Recruitment Feasibility (Eligibility) | One year from when the study starts enrolling participants
  The proportion of participants eligible to participate in Mother Matters

SECONDARY OUTCOMES:
Edinburgh Postnatal Depressive Scale (EPDS) | Follow-up (10 weeks post-randomization at the completion of the Mother Matters online support group for the immediate treatment condition arm)
  The investigators will measure depressive symptoms using the EPDS, a self-report depression screening measure that has been validated for use in pregnancy. EPDS scores >12 are predictive of a diagnosis of major depressive disorder.
State-Trait Anxiety Inventory (STAI) | Follow-up (10 weeks post-randomization at the completion of the Mother Matters online support group for the immediate treatment condition arm)
  The investigators will measure anxious symptoms using the STAI, a self-report anxiety screening measure that has shown good discriminate validity in perinatal populations. STAI scores >48 are predictive of having an anxiety disorder diagnosis.
The Change in Eating Disorder Symptoms Scale (CHEDS) | Follow-up (10 weeks post-randomization at the completion of the Mother Matters online support group for the immediate treatment condition arm)
  The investigators will measure eating disorder symptoms use the CHEDS, which is designed to assess change in eating disorder symptoms and their severity.
Parenting Stress Index, Short Form (PSI) | Follow-up (10 weeks post-randomization at the completion of the Mother Matters online support group for the immediate treatment condition arm)
  The investigators will measure stress in the parent-child relationship using the PSI short form, a 36-item measure which consists of three sub-scales.
Intervention Acceptability (Qualitative) | Follow-up (Immediate treatment condiction: 10 weeks post-randomization, i.e. at completion of the Mother Matters online support group; Waitlist control condition: 10 weeks after the waitlist Mother Matters group starts)
  Mother Matters Program Evaluation Questionnaire. This is comprised of open- and closed-ended questions to elicit feedback on a) content, clarity and helpfulness of the group, b) acceptability of the group format, c) satisfaction with the group, including reasons for discontinuation, d) the facilitators availability and helpfulness, and e) whether or not participants would recommend it to other women experiencing depressive symptoms in the first postpartum year.
Intervention Acceptability (Website Usage) | Follow-up (Immediate treatment condiction: 10 weeks post-randomization, i.e. at completion of the Mother Matters online support group; Waitlist control condition: 10 weeks after the waitlist Mother Matters group starts)
  Proportion of intervention weeks that participant logs in to the forum
Trial Protocol Adherence (Study Measure Completion) | Follow-up (about 10 weeks post-randomization)
  Proportion of participants who complete follow-up measures
Recruitment Feasibility (Recruitment) | One year from when the study starts enrolling participants
  The number of women recruited to the study
Trial Protocol Adherence (Weekly Posting) | Follow-up (Immediate treatment condiction: 10 weeks post-randomization, i.e. at completion of the Mother Matters online support group; Waitlist control condition: 10 weeks after the waitlist Mother Matters group starts)
  The number of participants who post in the forum at least on a weekly basis
Trial Protocol Adherence (Posting Drop-Off) | Follow-up (Immediate treatment condiction: 10 weeks post-randomization, i.e. at completion of the Mother Matters online support group; Waitlist control condition: 10 weeks after the waitlist Mother Matters group starts)
  The drop-off rate for postings (i.e. the number of participants who post in the initial weeks but not in the latter half of the group)

CONTACTS AND LOCATIONS:
Overall Officials: Simone Vigod, MD,MSc,FRCPC, Principal Investigator — Women's College Hospital
Locations (1):
- Women's College Research Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maternal depression and child development. Paediatr Child Health. 2004 Oct;9(8):575-598. doi: 10.1093/pch/9.8.575. No abstract available. PMID 19680490
- [Background] Marcus SM. Depression during pregnancy: rates, risks and consequences--Motherisk Update 2008. Can J Clin Pharmacol. 2009 Winter;16(1):e15-22. Epub 2009 Jan 22. PMID 19164843
- [Background] Meltzer-Brody S, Jones I. Optimizing the treatment of mood disorders in the perinatal period. Dialogues Clin Neurosci. 2015 Jun;17(2):207-18. doi: 10.31887/DCNS.2015.17.2/smeltzerbrody. PMID 26246794
- [Background] Roberta Anniverno, A.B., Claudio Mencacci and Federico Durbano, Anxiety Disorders in Pregnancy and the Postpartum Period, in New Insights into Anxiety Disorders, D.F. Durbano, Editor. 2013.
- [Background] Misri S, Abizadeh J, Sanders S, Swift E. Perinatal Generalized Anxiety Disorder: Assessment and Treatment. J Womens Health (Larchmt). 2015 Sep;24(9):762-70. doi: 10.1089/jwh.2014.5150. Epub 2015 Jun 30. PMID 26125602
- [Background] Farr SL, Dietz PM, O'Hara MW, Burley K, Ko JY. Postpartum anxiety and comorbid depression in a population-based sample of women. J Womens Health (Larchmt). 2014 Feb;23(2):120-8. doi: 10.1089/jwh.2013.4438. Epub 2013 Oct 26. PMID 24160774
- [Background] Easter A, Solmi F, Bye A, Taborelli E, Corfield F, Schmidt U, Treasure J, Micali N. Antenatal and postnatal psychopathology among women with current and past eating disorders: longitudinal patterns. Eur Eat Disord Rev. 2015 Jan;23(1):19-27. doi: 10.1002/erv.2328. Epub 2014 Oct 26. PMID 25345371
- [Background] Micali N, Simonoff E, Treasure J. Pregnancy and post-partum depression and anxiety in a longitudinal general population cohort: the effect of eating disorders and past depression. J Affect Disord. 2011 Jun;131(1-3):150-7. doi: 10.1016/j.jad.2010.09.034. Epub 2010 Dec 10. PMID 21146231
- [Background] Dennis CL, Chung-Lee L. Postpartum depression help-seeking barriers and maternal treatment preferences: a qualitative systematic review. Birth. 2006 Dec;33(4):323-31. doi: 10.1111/j.1523-536X.2006.00130.x. PMID 17150072
- [Background] Paul IM, Downs DS, Schaefer EW, Beiler JS, Weisman CS. Postpartum anxiety and maternal-infant health outcomes. Pediatrics. 2013 Apr;131(4):e1218-24. doi: 10.1542/peds.2012-2147. Epub 2013 Mar 4. PMID 23460682
- [Background] Yelland J, Sutherland G, Brown SJ. Postpartum anxiety, depression and social health: findings from a population-based survey of Australian women. BMC Public Health. 2010 Dec 20;10:771. doi: 10.1186/1471-2458-10-771. PMID 21167078
- [Background] National Collaborating Centre for Mental Health (UK). Antenatal and Postnatal Mental Health: Clinical Management and Service Guidance: Updated edition. Leicester (UK): British Psychological Society; 2014 Dec. Available from http://www.ncbi.nlm.nih.gov/books/NBK305023/ PMID 26180865
- [Background] Evans M, Donelle L, Hume-Loveland L. Social support and online postpartum depression discussion groups: a content analysis. Patient Educ Couns. 2012 Jun;87(3):405-10. doi: 10.1016/j.pec.2011.09.011. Epub 2011 Oct 20. PMID 22019021
- [Background] Spangler DL. The Change in Eating Disorder Symptoms scale: scale development and psychometric properties. Eat Behav. 2010 Aug;11(3):131-7. doi: 10.1016/j.eatbeh.2009.12.003. Epub 2009 Dec 11. PMID 20434058
- [Background] Haskett ME, Ahern LS, Ward CS, Allaire JC. Factor structure and validity of the parenting stress index-short form. J Clin Child Adolesc Psychol. 2006 Jun;35(2):302-12. doi: 10.1207/s15374424jccp3502_14. PMID 16597226
- [Background] Harris AA. Practical advice for caring for women with eating disorders during the perinatal period. J Midwifery Womens Health. 2010 Nov-Dec;55(6):579-86. doi: 10.1016/j.jmwh.2010.07.008. PMID 20974420
- [Background] Micali N, Simonoff E, Stahl D, Treasure J. Maternal eating disorders and infant feeding difficulties: maternal and child mediators in a longitudinal general population study. J Child Psychol Psychiatry. 2011 Jul;52(7):800-7. doi: 10.1111/j.1469-7610.2010.02341.x. Epub 2010 Nov 12. PMID 21073463
- [Background] Coker E, Abraham S. Body weight dissatisfaction before, during and after pregnancy: a comparison of women with and without eating disorders. Eat Weight Disord. 2015 Mar;20(1):71-9. doi: 10.1007/s40519-014-0133-4. Epub 2014 Jun 7. PMID 24906550
- [Background] Hertzog MA. Considerations in determining sample size for pilot studies. Res Nurs Health. 2008 Apr;31(2):180-91. doi: 10.1002/nur.20247. PMID 18183564
- [Background] Meltzer-Brody S, Zerwas S, Leserman J, Holle AV, Regis T, Bulik C. Eating disorders and trauma history in women with perinatal depression. J Womens Health (Larchmt). 2011 Jun;20(6):863-70. doi: 10.1089/jwh.2010.2360. PMID 21671774